CLINICAL TRIAL: NCT01398917
Title: Multicenter Randomized Trial Comparing Short-term Stenting Versus Balloon Dilatation for Dominant Strictures in Primary Sclerosing Cholangitis
Brief Title: Short-term Stenting Versus Balloon Dilatation for Dominant Strictures in Primary Sclerosing Cholangitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, C.Y. Ponsioen, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DILSTENT2; NL34454.018.10 (Registry Identifier: CCMO, Netherlands)
Record Dates: First submitted 2011-04-25; First posted 2011-07-21 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: psc; dominant stricture
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- short-term stenting (Active Comparator): one 10 Fr Plastic endoprosthesis or 2 7 Fr plastic endoprosthesis inserted through dominant stricture(s), to be extracted after 1-2 weeks
  Interventions: Procedure: plastic endoprosthesis
- balloon dilatation (Active Comparator): 4 cm 6 mm biliary dilatation balloon to be inflated for 2 minutes in dominant stricture(s)
  Interventions: Procedure: balloon dilatation

INTERVENTIONS:
Procedure: plastic endoprosthesis — one 10 Fr Plastic endoprosthesis or 2 7 Fr plastic endoprosthesis inserted through dominant stricture(s), to be extracted after 1-2 weeks
  Other Names: plastic stent
  Arms: short-term stenting
Procedure: balloon dilatation — 4 cm 6 mm biliary dilatation balloon to be inflated for 2 minutes in dominant stricture(s)
  Other Names: biliary dilatation balloon
  Arms: balloon dilatation

SUMMARY:
Primary sclerosing cholangitis (PSC) is a chronic inflammatory disease of the biliary tract of unknown origin. Around 50% of patients develop during their disease course narrowing of the main bile duct with corresponding increase in symptoms such as itching, jaundice and abdominal pain. These narrowings can be treated by balloon dilatation or temporary insertion of a plastic endoprosthesis. However, it is not known which of these two therapeutic modalities is best. This study aims to compare both techniques in order to determine which is best in terms of postponing recurrence of the narrowing, safety and costs.

DETAILED DESCRIPTION:
Rationale:

Primary sclerosing cholangitis is a chronic progressive fibro-obliterative disease of the biliary tree leading to biliary cirrhosis. During its course, dominant strictures occur in approximately 50% of patients. These can be accompanied by lead worsening of symptoms and jaundice and are an indication for endoscopic treatment. The best form of treatment, either balloon dilatation or short-term stent placement, has never been formally investigated.

Objective:

Primary:

To compare the efficacy of single session balloon dilatation versus short-term stent placement in non-advanced PSC patients with regard to re-intervention free recurrence rate at two years.

Secondary:

To compare the short term efficacy of single balloon dilatation versus short-term stenting with regard to improvement of cholestatic symptoms, biochemical cholestasis, and quality of life in non-endstage PSC patients at three months; to compare the safety of single balloon dilatation session versus short-term stenting in non advanced PSC patients during two years.

Study design: This is a multicenter, open-label, randomized intervention study.

Study population:

Non-advanced primary sclerosing cholangitis subjects with progression of cholestatic complaints from the outpatient population of the seven participating centres.

Main study parameters/endpoints:

1. Difference in re-intervention free survival time between both groups at two years.
2. Change in semi-quantitative scoring of cholestatic symptoms (pruritus, right upper quadrant pain, fatigue) from baseline at three months.
3. Change in total bilirubin, alkaline phosphatase, and yGT from baseline at 3 months.
4. Safety: adverse events, clinical laboratory values, vital signs.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Currently, both interventions belong to standard patient care armamentarium. Burden for the patient exists in slightly more regular follow-up visits for two years (three-monthly instead of every 3-4 months) to their treating centre. ERCP is associated with a low mortality (<0.5 %) and acceptable morbidity (overall 5%). Most dreaded complications are severe post-ERCP pancreatitis (<2%) and suppurative cholangitis (<2%). From the available retrospective literature data the incidence of these complications does not seem to differ between the two treatment modalities. ERCP will only be performed when there is a clearcut clinical indication anyway.

ELIGIBILITY:
Inclusion Criteria:

* PSC ascertained with MRCP, ERCP, PTC and/or liver biopsy or
* PSC highly suspected and to be confirmed with present ERCP
* Age between 18-75 years
* Total bilirubin > 3x ULN or rsie in alkaline phosphatase or bilirubin > 50% together with increase in cholestatic complaints

Exclusion Criteria:

* Prior stenting or balloon-dilatation within last 6 months
* Clinical signs serious suppurative cholangitis reflected by either fever > 39.0 °C, tachycardia, leukocytosis and elevated CRP, or fever > 38,5 C together with purulent bile found during ERCP.
* Change of ursodeoxycholic acid therapy shorter than two months ago.
* Inability to give written informed consent
* Signs of biliary cirrhosis Child-Pugh B or C
* Estimated transplant-free survival shorter than 2 years as calculated by a Mayo score < 2
* Serious suspicion of cholangiocarcinoma, reflected by an imaging study suggestive of metastasis, MRCP with mass lesion with contrast enhancement, rise in CA19.9 of > 63 U/ml with an absolute value > 130 U/ml 14 .
* Signs of current malignancy other than basocellular skin carcinoma.
* Inability to give informed consent.
* Life expectancy < 24 months.
* Use of antibiotics in previous 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
recurrence-free interval of the primary dominant stricture | 24 months

SECONDARY OUTCOMES:
number of patients with adverse events in both groups | 3 months
  adverse events within first 3 months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Cyriel Y Ponsioen, dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (4):
- UZLeuven, Leuven, Belgium
- Academic Medical Center, Amsterdam, Netherlands
- Rikshospitalet, Oslo, Norway
- Karolinska Institute, Stockholm, Sweden

REFERENCES:
- [Derived] Ponsioen CY, Arnelo U, Bergquist A, Rauws EA, Paulsen V, Cantu P, Parzanese I, De Vries EM, van Munster KN, Said K, Chazouilleres O, Desaint B, Kemgang A, Farkkila M, Van der Merwe S, Van Steenbergen W, Marschall HU, Stotzer PO, Thorburn D, Pereira SP, Aabakken L. No Superiority of Stents vs Balloon Dilatation for Dominant Strictures in Patients With Primary Sclerosing Cholangitis. Gastroenterology. 2018 Sep;155(3):752-759.e5. doi: 10.1053/j.gastro.2018.05.034. Epub 2018 May 24. PMID 29803836